CLINICAL TRIAL: NCT00394251
Title: An Open-label, Randomized, Comparative Pilot Study of Dose-dense Adriamycin Plus Cytoxan (AC) Followed by Either ABI-007 (Abraxane) or Taxol With Bevacizumab as Adjuvant Therapy for Patients With Breast Cancer
Brief Title: Study of Dose-dense Adriamycin Plus Cytoxan (AC) Followed by Either ABI-007 (Abraxane) or Taxol With Bevacizumab as Adjuvant Therapy for Patients With Breast Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Celgene (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CA045
Record Dates: First submitted 2006-10-30; First posted 2006-10-31 (Estimated); Results first posted 2013-07-18 (Estimated); Last update posted 2019-11-25 (Actual); Status verified 2019-11

CONDITIONS: Breast Cancer
Keywords: Adjuvant therapy; Bevacizumab; Abraxane; Early stage breast cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Doxorubicin; Cyclophosphamide; Albumin-Bound Paclitaxel; Paclitaxel; Bevacizumab; pegfilgrastim

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- AC --> ABI-007 (Experimental): Adriamycin and Cytoxan plus Bevacizumab for four cycles (weeks 1-8); 260 mg/m^2 ABI-007 (Abraxane) plus Bevacizumab for four cycles (weeks 9-16); Bevacizumab (weeks 17-46).
  Interventions: Drug: Adriamycin and Cytoxan (AC); Drug: ABI-007; Drug: Bevacizumab; Drug: pegfilgrastim
- AC --> Taxol (Experimental): Adriamycin and Cytoxan plus Bevacizumab for four cycles (weeks 1-8); 175 mg/m^2 Taxol plus Bevacizumab for four cycles (weeks 9-16); Bevacizumab (weeks 17-46).
  Interventions: Drug: Adriamycin and Cytoxan (AC); Drug: Taxol; Drug: Bevacizumab; Drug: pegfilgrastim

INTERVENTIONS:
Drug: Adriamycin and Cytoxan (AC) — Adriamycin (doxorubicin) and Cytoxan (cyclophosphamide) make up the chemotherapy regimen known as AC. Adriamycin 60 mg/m^2 intravenous, plus Cytoxan 600 mg/m^2 intravenous on Day 1 of each of four 2-week cycles (weeks 1-8).
  Other Names: doxorubicin; cyclophosphamide
Drug: ABI-007 — 260 mg/m^2 IV on day 1 of each of four 2-week cycle, representing treatment cycles 5-8 (weeks 9-16)
  Other Names: Abraxane
  Arms: AC --> ABI-007
Drug: Taxol — 175 mg/m^2 intravenously (IV) on day 1 of each of four 2-week cycle, representing treatment cycles 5-8 (weeks 9-16)
  Other Names: paclitaxel
  Arms: AC --> Taxol
Drug: Bevacizumab — 10 mg/kg on day 1 of each of eight 2-week cycles (weeks 9-16), then 15 mg/kg on day 1 of each of ten three-week cycles (weeks 17-46).
  Other Names: Avastin®
Drug: pegfilgrastim — 6 mg subcutaneous (SC) on day 2 for each of the first four 2-week cycles (weeks 1-8). Pegfilgrastim 6 mg SC was administered on day 2 of cycles 6-8 (weeks 11-16) during taxane treatment only if necessary.
  Other Names: Neulasta

SUMMARY:
The primary objective of this study was to compare the safety of dose-dense ABI-007 (Abraxane) 260 mg/m^2 or Taxol 175 mg/m^2 given every 2 weeks following dose-dense Adriamycin plus Cytoxan (AC) chemotherapy. Bevacizumab was administered at 10 mg/kg every 2 weeks throughout chemotherapy, and then at 15 mg/kg every 3 weeks following chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

A patient was eligible for inclusion in this study only if all of the following criteria were met:

1. Female, age greater than or equal to 18 to less than or equal to 70 years old.
2. Estrogen receptor (ER) and progesterone receptor (PR) status have been determined.
3. Operable, histologically confirmed adenocarcinoma of the breast
4. Must have met 1 of the following criteria:

   * T1-3, N1-3, M0, regardless of ER or PR status.
   * T > 2 cm, N0, M0 (T2-3N0M0), regardless of ER or PR status.
   * T > 1 cm, N0, M0 (T1cN0M0) and both ER and PR negative
   * T > 1 cm, N0, M0, ER or PR positive and grade 3
5. Patients with one sentinel lymph node metastasis 0.2-2 mm in size were not required to undergo completion axillary dissection unless only 1 sentinel lymph node was examined. This completion axillary dissection was optional if 1 out of 2 or more sentinel lymph nodes was positive for a micrometastasis. Therefore if 1 of 1 sentinel lymph node was positive for micrometastasis(0.2-2 mm), then a completion axillary dissection was required.
6. Patients with more than one sentinel node micrometastasis or 1 node with a micrometastasis > 2 mm and/or T3 disease must have undergone completion, standard axillary dissection. -Note: the following were not eligible-

   T1b,c,N0M0 and ER or PR positive and grade 1 or 2 Tx tumors (regardless of nodal status) T4 disease [i.e., patients with fixed tumors, peau d'orange skin changes, skin ulcerations, or inflammatory changes
   * Note: Sentinel lymph node micrometastasis < 0.2 mm in considered N0 disease
7. Negative surgical margins on lumpectomy or mastectomy specimen (no ink on invasive cancer and no ink on ductal carcinoma in situ [DCIS]).
8. Eastern Cooperative Oncology Group (ECOG) performance status 0-1
9. Normal electrocardiogram (ECG, as assessed by the investigator).
10. No pre-existing peripheral neuropathy.
11. It had not been longer than 84 days since the date of definitive surgery (eg, mastectomy or in the case of a breast-sparing procedure, axillary dissection).
12. Laboratory values were to be as follows:

    * White blood cell count: > or equal to 3,000/mm^3
    * Absolute neutrophil count:> or equal to 1,500/mm^3
    * Platelets:> or equal to 100,000/mm^3
    * Hemoglobin: > or equal to 8g/dL
    * Bilirubin:< or equal to the institution's ULN
    * Creatinine: < or equal to 1.7 mg/dL
    * Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) and alkaline phosphatase could be up to 2.5 times the institutional ULN.
13. All staging studies including physical exam, chest x-ray, and bone scan had to show no evidence of metastatic disease, including suspicious lymphadenopathy or skin nodules on physical exam. A chest x-ray and bone scan were mandatory; however, all other staging studies were at the treating physician's discretion. Any other staging test (eg, Computed Tomography [CT] scans, magnetic resonance imaging [MRI] studies, ultrasound of abdomen, Positron Emission Tomography [PET] scans must have been negative for metastatic disease. An abdominal CT scan or PET scan was mandatory for patients with liver function tests elevated above the upper limit of normal (ULN) to rule out metastatic disease. If the patient had a staging PET scan then a bone scan was not necessary, but a chest x-ray was required.
14. Patient had a negative serum pregnancy test < or equal to 14 days of the first dose of study drug (patients of childbearing potential).
15. If fertile, patient had agreed to us an acceptable method of birth control to avoid pregnancy [Note: oral contraceptives were not allowed] for the duration of chemotherapy and hormonal therapy and for 6 months thereafter.
16. If obese, a patient must have been treated with doses calculated using his/her actual body surface area (BSA) (the physician must have been comfortable treating at the full BSA dose regardless of BSA).
17. Patient had signed a Patient Informed Consent Form.

Exclusion Criteria:

A patient was not eligible for inclusion in this study if any of the following criteria applied:

1. Patients with HER-2 positive breast cancer (IHC 3+ or FISH +) who were eligible for adjuvant Herceptin therapy.
2. Stage IV breast cancer (M1 disease on TNM staging system).
3. Prior anthracycline, anthracenedione (mitoxantrone), or taxane therapy
4. Neoadjuvant therapy for this breast cancer.
5. Previous invasive cancers if treated < 5 years prior to entering this study, except basal or squamous cell carcinoma of the skin or carcinoma in situ of the cervix; the latter were not required to have occurred more than 5 years prior to study entry.
6. Prior invasive breast cancer if diagnosed < 5 years prior to entering study. Patients must have finished adjuvant hormonal therapy prior to registration. Patients with prior DCIS are eligible. Patients with DCIS who were treated with tamoxifen must have finished tamoxifen prior to registration.
7. Serious medical illness, other than that treated by this study, which would limit survival to < 4 years, or psychiatric condition that would prevent informed consent and compliance with study treatment.
8. Uncontrolled or severe cardiovascular disease including recent (< or equal to 12 months) myocardial infarction or unstable angina.
9. Active uncontrolled bacterial, viral (including clinically defined Acquired Immune Deficiency Syndrome [AIDS]), or fungal infection.
10. Patients with active or chronic hepatitis with abnormal liver function tests (LFTs) or patients who were known to be HIV positive.
11. Uncontrolled disease such as uncontrolled diabetes.
12. Any prior history of hypertensive crisis or hypertensive encephalopathy.
13. Any known central nervous system (CNS) disease.
14. Known hypersensitivity to any component of bevacizumab.
15. No history of cerebrovascular accident or transient ischemic attack at any time.
16. Active symptomatic vascular disease, e.g., aortic aneurysm or aortic dissection, and no peripheral vascular disease, e.g., claudication, within six months of study entry.
17. No major surgical procedure, open biopsy, or significant traumatic injury within 28 days and no core biopsy or minor surgical procedure (excluding placement of a vascular access device) within seven days of study entry. No anticipated need for major surgical procedure during the course of study.
18. No history of abdominal fistula, gastrointestinal perforation, or intra- abdominal process within six months of study entry.
19. No serious non-healing wound, ulcer, or bone fracture.
20. No proteinuria at screening as demonstrated by urine protein: urine creatinine (UPC) ratio of > or equal to 1.0 or urine dipstick for proteinuria > or equal to 2+ (patients discovered to have > or equal to 2+ proteinuria on dipstick urinalysis at baseline should have undergone a 24 hour urine collection and must have demonstrated < or equal to 1g of protein in 24 hours to be eligible).
21. Inadequately controlled hypertension (defined as systolic blood pressure > 150 mmHg and /or diastolic blood pressure> 100 mmHg on antihypertensive medications) or New York Heart Association (NYHA) Grade 2 or greater congestive heart failure.
22. History or coagulopathy, bleeding diathesis, therapeutic anticoagulation other than low dose or chronic acetyl salicylic acid (ASA)> or equal to 325 mg. per day. Low dose coumadin for anticoagulation of venous access device or low dose molecular weight heparin (LMWH) for deep vein thrombosis prophylaxis or low dose (325 mg or less) ASA prophylaxis are allowed, but are best avoided if the treating physician feels it is safe to do so.
23. Left Ventricular Ejection Fraction (LVEF) on cardiac echocardiography (ECHO) < 50% (or institutional lower limit of normal [LLN]) and > or equal to 74%. LVEF of greater than 75% at baseline should have been re- reviewed and/or the test repeated as it could be falsely elevated.
24. Patients who were receiving concurrent immunotherapy.
25. A history of other malignancy within the last 5 years, which could affect the diagnosis or assessment of breast cancer recurrence or which could shorten a patient's survival.
26. Patient had had an organ allograft.
27. Patient was pregnant or breastfeeding.
28. Patient was unable to comply with requirements of study.
29. Patient was receiving any other investigational drugs.

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 197 (Actual)
Dates: Start 2006-08-01 (Actual); Primary Completion 2007-03-01 (Actual); Study Completion 2008-02-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (26):
- United States (26):
  - Birmingham, Alabama
  - Sedona, Arizona
  - Denver, Colorado
  - Torrington, Connecticut
  - Indianapolis, Indiana
  - Minneapolis, Minnesota
  - Columbia, Missouri
  - St Louis, Missouri
  - Henderson, Nevada
  - Raleigh, North Carolina
  - Eugene, Oregon
  - Greenville, South Carolina
  - Austin, Texas
  - Bedford, Texas
  - Dallas, Texas
  - El Paso, Texas
  - Fort Worth, Texas
  - Fredericksburg, Texas
  - Houston, Texas
  - Longview, Texas
  - McAllen, Texas
  - Tyler, Texas
  - Waco, Texas
  - Fairfax, Virginia
  - Norfolk, Virginia
  - Vancouver, Washington

REFERENCES:
- [Result] Pippen J, Paul D, Vukelja S, Clawson A, Iglesias J. Dose-dense doxorubicin and cyclophosphamide followed by dose-dense albumin-bound paclitaxel plus bevacizumab is safe as adjuvant therapy in patients with early stage breast cancer. Breast Cancer Res Treat. 2011 Dec;130(3):825-31. doi: 10.1007/s10549-011-1678-9. Epub 2011 Oct 6. PMID 21976055

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Multicenter study
Pre-assignment Details: Two hundred three patients were randomized and one hundred ninety-seven were treated.
Period: Overall Study
Arm/Group | AC --> ABI-007 | AC --> Taxol
Started | 98 | 99
At Least One Dose of Taxane | 93 | 93
Completed | 61 | 61
Not Completed | 37 | 38
Not completed — Adverse Event | 7 | 5
Not completed — Unacceptable Toxicity | 20 | 18
Not completed — Physician Decision | 1 | 1
Not completed — Protocol Violation | 0 | 1
Not completed — Withdrawal by Subject | 7 | 11
Not completed — Non-compliance, pt moved, pt/inv agree | 2 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | AC --> ABI-007 | AC --> Taxol | Total
Number analyzed (Participants) | 98 | 99 | 197
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.2 (9.21) | 51.2 (9.29) | 51.2 (9.23)
Age, Customized [Number; unit: participants]
  >=65 years | 9 | 11 | 20
  < 65 years | 89 | 88 | 177
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 98 | 99 | 197
  Male | 0 | 0 | 0
Race/Ethnicity, Customized [Number; unit: participants]
  Asian | 3 | 2 | 5
  White, non-Hispanic, non-Latino | 76 | 72 | 148
  White, Hispanic or Latino | 8 | 17 | 25
  Black, of African heritage | 10 | 7 | 17
  Other | 1 | 1 | 2
Region of Enrollment [Number; unit: participants]
  United States | 98 | 99 | 197
Weight [Mean (Standard Deviation); unit: kg] | 78.63 (19.561) | 78.78 (19.595) | 78.71 (19.528)
Menopausal Status [Number; unit: participants]
  premenopausal | 50 | 44 | 94
  postmenopausal | 48 | 55 | 103
Stage at Primary Diagnosis [Number; unit: participants] — American Joint Committee on Cancer (AJCC) 6th edition staging for breast cancer was used to define stage at primary diagnosis. The scale ranges from stage I (primary tumor <=2.0 cm, no regional or distant lymph node involvement) to stage IV (primary tumor of any size, with both regional and distant lymph node involvement). Each stage includes combinations of ratings for the primary tumor, regional lymph node involvement, and metastasis. Illustrative examples of stages appear in the data table. Each higher stage represents increasingly poor prognosis.
  participants
    I: tumor <=2.0, lymph nodes clear, no metastasis | 10 | 7 | 17
    IIa: tumor <=2.0 cm, regional lymph node | 28 | 35 | 63
    IIb: tumor >2.0<5.0cm, regional lymph nodes | 32 | 24 | 56
    IIIa: tumor may be >5.0 cm, regional lymph nodes | 22 | 23 | 45
    IIIb: tumor extending to chest wall or skin | 0 | 0 | 0
    IIIc: tumor with extensive lymph node involvement | 6 | 9 | 15
    IV: distant metastasis | 0 | 0 | 0
    unknown | 0 | 1 | 1
Estrogen Receptor Status [Number; unit: participants] — Defined as detectable presence (positive) or absence (negative) of estrogen receptors in tumor biopsy sample
  participants
    Positive | 63 | 66 | 129
    Negative | 35 | 33 | 68
Progesterone Receptor Status [Number; unit: participants] — Defined as detectable presence (positive) or absence (negative) of progesterone receptors in tumor biopsy sample
  participants
    Positive | 59 | 59 | 118
    Negative | 39 | 40 | 79
Eastern Cooperative Oncology Group (ECOG) Performance Status [Number; unit: participants] — Using Eastern Cooperative Oncology Group (ECOG) performance status scale (Oken, M.M., Creech, R.H., Tormey, D.C., Horton, J., Davis, T.E., McFadden, E.T., Carbone, P.P.: Toxicity And Response Criteria Of The Eastern Cooperative Oncology Group. Am J Clin Oncol 5:649-655, 1982).
  participants
    0 (Fully active) | 89 | 89 | 178
    1 (Restrictive but ambulatory) | 9 | 10 | 19
Physician's Assessment of Peripheral Neuropathy [Number; unit: participants] — Physician's evaluation of peripheral neuropathy used the National Cancer Institute's Common Terminology Criteria for Adverse Events v3.0 (NCI CTCAE Version 3.0) severity scale which is a five step scale with 1=mild adverse event and 5 = death related to an adverse event.
  participants
    0 (None) | 94 | 96 | 190
    1 | 1 | 0 | 1
    Not reported | 3 | 3 | 6

OUTCOME MEASURES:

1. Secondary Outcome: The Cumulative Dose of Taxane Delivered During Study
Description: The cumulative dose of taxane (Taxol or ABI-007) taken during the study (cycles 4-8 which is approximately weeks 9-16).
Time Frame: approximately week 9-16
Population: Participants in the treated population who received at least 1 dose of taxane.
Measure: Mean (Standard Deviation); unit: mg/m^2
Arm/Group | AC --> ABI-007 | AC --> Taxol
Number analyzed (Participants) | 93 | 93
mg/m^2 | 950.5 (199.86) | 660.8 (99.52)

2. Secondary Outcome: Mean Taxane Dose Intensity Per Week
Description: Cumulative taxane (ABI-007 or Taxol) dose divided by the number of weeks on taxane treatment.
Time Frame: approximately week 9-16
Population: Participants in the treated population who received at least 1 dose of taxane.
Measure: Mean (Standard Deviation); unit: mg/m^2/week
Arm/Group | AC --> ABI-007 | AC --> Taxol
Number analyzed (Participants) | 93 | 93
mg/m^2/week | 118.82 (24.983) | 82.60 (12.440)

3. Primary Outcome: Participants With Treatment-Emergent Toxicities With a Frequency >=20% at 3 Months Post Chemotherapy
Description: Toxicities are summarized using the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) terms. Participants with treatment-emergent toxicities with a frequency of >=20% in any treatment arm, and participants with at least one toxicity are reported.
  Taxane subsets (ABI-007 subset and Taxol subset treatment arms) summarize participants with treatment-emergent toxicities defined as any AEs that begin or worsen in severity grade after the start of taxane treatment (cycle 5, week 9) through 30 days after the last dose of taxane (week 20) and were ongoing 3 months after chemotherapy (month 7).
  Entire regiments (AC --> ABI-007 and AC --> Taxol treatment arms) summarize participants with treatment-emergent toxicities defined as any AEs that begin or worsen in severity grade after the start of chemotherapy (cycle 1, week 1) through 30 days after the last dose of chemotherapy (week 20) and were ongoing 3 months after chemotherapy (month 7).
Time Frame: Month 7
Population: Participants in the Treated Population for whom safety data was available 3 months post-chemotherapy
Measure: Number; unit: participants
Groups:
- ABI-007 Subset: 260 mg/m2 ABI-007 (Abraxane) plus Bevacizumab for 4 cycles (weeks 9-16); Bevacizumab (weeks 17-46). Weeks 1-8 are excluded from this subset.
- AC --> ABI-007: Adriamycin and Cytoxan plus Bevacizumab for four cycles (weeks 1-8); 260 mg/m2 ABI-007 (Abraxane) plus Bevacizumab for 4 cycles (weeks 9-16); Bevacizumab (weeks 17-46).
- Taxol Subset: 175 mg/m2 Taxol plus Bevacizumab for 4 cycles (weeks 9-16); Bevacizumab (weeks 17-46). Weeks 1-8 are excluded from this subset.
- AC --> Taxol: Adriamycin and Cytoxan plus Bevacizumab for four cycles (weeks 1-8); 175 mg/m2 Taxol plus Bevacizumab for 4 cycles (weeks 9-16); Bevacizumab (weeks 17-46).
Arm/Group | ABI-007 Subset | AC --> ABI-007 | Taxol Subset | AC --> Taxol
Number analyzed (Participants) | 74 | 74 | 77 | 77
participants
  At least 1 AE at 3 Months | 65 | 74 | 65 | 77
  Neurology: Neuropathy: Sensory | 36 | 50 | 28 | 35
  Constitutional Symptoms: Fatigue | 16 | 46 | 10 | 32
  Dermatology/Skin: Hair Loss/Alopecia (Scalp+Body) | 2 | 33 | 1 | 17
  Endocrine: Hot Flashes/Flushes | 12 | 28 | 5 | 22
  Cardiac General: Hypertension | 4 | 18 | 7 | 25
  Pain: Arthralgia | 7 | 22 | 8 | 19
  Hemorrhage/Bleeding: Nasal | 11 | 19 | 10 | 18
  Pain: Other - Extremity | 4 | 15 | 7 | 22
  Pain: Myalgia | 10 | 20 | 9 | 16
  Dermatology/Skin: Nail Changes | 14 | 22 | 5 | 10
  Constitutional Symptoms: Insomnia | 3 | 16 | 5 | 11
Statistical Analysis 1: Comparison: ABI-007 Subset vs Taxol Subset; Comparison of percentage of participants with at least one taxane-emergent toxicity; Test type: Superiority or Other; p = 0.641, Fisher Exact

4. Secondary Outcome: Percent of Protocol Taxane Dose
Description: Percent of the protocol-defined taxane (ABI-007 or Taxol) dose that was actually taken by study participants.
Time Frame: approximately week 9-16
Population: Participants in the treated population who received at least 1 dose of taxane.
Measure: Mean (Standard Deviation); unit: percentage of protocol-defined taxane
Arm/Group | AC --> ABI-007 | AC --> Taxol
Number analyzed (Participants) | 93 | 93
percentage of protocol-defined taxane | 91.40 (19.218) | 94.40 (14.217)

5. Secondary Outcome: Summary of Participant Treatment Exposure, Dose Interruptions, Dose Reductions, and Dose Delays
Description: Counts of participants who
  * completed the protocol-defined treatment cycles,
  * had a dose interruption
  * had a dose reduction
  * had a dose delay. A dose delay refers to the delay of all interventions in the cycle.
  Dose modifications are typically caused by clinically significant laboratory abnormalities and /or treatment emergent adverse events/toxicities.
  Use of pegfilgrastim is included in the summary.
Time Frame: up to Week 46
Population: Treated population
Measure: Number; unit: participants
Arm/Group | AC --> ABI-007 | AC --> Taxol
Number analyzed (Participants) | 98 | 99
participants
  Completed 4 cycles of Adriamycin/Cytoxan (AC) | 95 | 95
  Received pegfilgrastim for 4 cycles during AC | 95 | 94
  Completed 4 cycles of taxane | 82 | 84
  Completed 18 cycles of bevacizumab | 61 | 61
  One or more dose reduction: Adriamycin | 10 | 6
  One or more dose reduction: Cytoxan | 9 | 5
  One or more dose reduction: Taxane | 12 | 16
  One or more dose interruption: Adriamycin | 1 | 0
  One or more dose interruption: Cytoxan | 3 | 1
  One or more dose interruption: Taxane | 0 | 3
  One or more dose interruption: Bevacizumab | 0 | 2
  One or more delay in study regimen | 50 | 48
  Discontinued pegfilgrastim during AC cycles | 0 | 0
  Administered pegfilgrastim during taxane cycles | 23 | 13

6. Secondary Outcome: Myelosuppression During Taxane Dosing Cycles
Description: Myelosuppression represented by neutropenia (low absolute neutrophil counts (ANC)) with severity grades according to Common Terminology Criteria for Adverse Events v3.0 (CTCAE).
  * Grade 1 = <lower limit of normal (LLN)-1.5*10^9/L
  * Grade 2 = <1.5 - 1.0*10^9/L
  * Grade 3 = <1.0 - 0.5*10^9/L
  * Grade 4 = <0.5*10^9/L
  Values are reported across all severity grades without assessment of relationship to taxane treatment, and also by relation to taxane treatment as reported by investigators.
Time Frame: Weeks 9-16
Population: Participants in the treated population who received at least 1 dose of taxane and had laboratory values.
Measure: Number; unit: participants
Arm/Group | AC --> ABI-007 | AC --> Taxol
Number analyzed (Participants) | 92 | 93
participants
  ANC (grades 1-4) | 58 | 43
  Taxane-related, grades 1-4 | 11 | 8
  Taxane-related, grades 3-4 | 6 | 5

7. Secondary Outcome: Change From Baseline in Percent Left Ventricular Ejection Fraction (% LVEF) at the Final Evaluation
Description: Decreased left ventricular ejection fraction (LVEF) is an indication of cardiotoxicity. Change from baseline measurements to the final evaluation are summarized.
Time Frame: up to week 46
Population: Participants in the treated population who had both baseline and one treatment measurement for %LVEF
Measure: Median (Full Range); unit: percentage of healthy LVEF
Arm/Group | AC --> ABI-007 | AC --> Taxol
Number analyzed (Participants) | 95 | 92
percentage of healthy LVEF | -1.0 (7.40) [-30 to 16] | -1.0 (93.40) [-699 to 16]

8. Secondary Outcome: Summary of Participants' Most Severe Grade for Liver and Renal Function Laboratory Adverse Experiences During Study (All Treatment Cycles)
Description: Summary of the most severe grades using the National Cancer Institute's Common Terminology Criteria for Adverse Events v3.0 (CTCAE) for the following liver and renal function tests.
  Grade 0 = within normal range for all measurements.
  Alkaline phosphatase, alanine aminotransferase (ALT), aspartate aminotransferase (AST):
  * Grade 1 = > upper limit of normal (ULN) - 2.5*ULN
  * Grade 2= >2.5-5.0*ULN
  * Grade 3= >5.0-20.0*ULN
  * Grade 4= >20.0*ULN
  Bilirubin:
  * Grade 1= >ULN - 1.5*ULN
  * Grade 3= >3.0 - 10.0*ULN
  Creatinine:
  - Grade 1= >ULN - 1.5*ULN
Time Frame: Week 1 up to week 50
Population: Treated population with at least one post-treatment laboratory measure.
Measure: Number; unit: participants
Arm/Group | AC --> ABI-007 | AC --> Taxol
Number analyzed (Participants) | 96 | 99
participants
  Alkaline phosphatase, Grade 0 | 69 | 70
  Alkaline phosphatase, Grade 1 | 26 | 29
  Alkaline phosphatase, Grade 2 | 1 | 0
  ALT, Grade 0 | 66 | 75
  ALT, Grade 1 | 24 | 23
  ALT, Grade 2 | 5 | 1
  ALT, Grade 4 | 1 | 0
  AST, grade 0 | 74 | 81
  AST, grade 1 | 20 | 17
  AST, grade 2 | 1 | 1
  AST, grade 3 | 1 | 0
  Bilirubin, grade 0 | 95 | 98
  Bilirubin, grade 1 | 0 | 1
  Bilirubin, grade 3 | 1 | 0
  Creatinine, grade 0 | 94 | 97
  Creatinine, grade 1 | 2 | 2

9. Primary Outcome: Participants With Treatment-Emergent Toxicities With a Frequency >=20% at 6 Months Post Chemotherapy
Description: Toxicities are summarized using the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) terms. Participants with treatment-emergent toxicities with a frequency of >=20% in any treatment arm, and participants with at least one toxicity are reported.
  Taxane subsets (ABI-007 subset and Taxol subset treatment arms) summarize participants with treatment-emergent toxicities defined as any AEs that begin or worsen in severity grade after the start of taxane treatment (cycle 5, week 9) through 30 days after the last dose of taxane (week 20) and were ongoing 6 months after chemotherapy (month 10).
  Entire regiments (AC --> ABI-007 and AC --> Taxol treatment arms) summarize participants with treatment-emergent toxicities defined as any AEs that begin or worsen in severity grade after the start of chemotherapy (cycle 1, week 1) through 30 days after the last dose of chemotherapy (week 20) and were ongoing 6 months after chemotherapy (month 10).
Time Frame: Month 10
Population: Participants in the Treated Population for whom safety data was available 6 months post-chemotherapy
Measure: Number; unit: participants
Arm/Group | ABI-007 Subset | AC --> ABI-007 | Taxol Subset | AC --> Taxol
Number analyzed (Participants) | 63 | 63 | 67 | 67
participants
  At least 1 AE at 6 Months | 49 | 62 | 46 | 65
  Neurology: Neuropathy: Sensory | 25 | 42 | 15 | 19
  Constitutional Symptoms: Fatigue | 11 | 32 | 4 | 18
  Endocrine: Hot Flashes/Flushes | 7 | 23 | 3 | 17
  Cardiac General: Hypertension | 4 | 12 | 7 | 18
  Pain: Arthralgia | 4 | 17 | 3 | 13
  Pain: Myalgia | 8 | 17 | 4 | 8
  Pain: Other - Extremity | 1 | 6 | 5 | 14
  Dermatology/Skin: Nail Changes | 8 | 13 | 3 | 6
Statistical Analysis 1: Comparison: ABI-007 Subset vs Taxol Subset; Comparison of percentage of participants with at least one taxane-emergent toxicity; Test type: Superiority or Other; p = 0.323, Fisher Exact

ADVERSE EVENTS:
Time Frame: Day 1 - up to week 50 (weeks 1-46 treatment, plus 30 days after last study dose)
Arm/Group | AC --> ABI-007 | AC --> Taxol
Serious Adverse Events (participants affected / at risk) | 30/98 | 21/99
Other Adverse Events (participants affected / at risk) | 97/98 | 99/99
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | AC --> ABI-007 (N=98) | AC --> Taxol (N=99)
Appendicitis perforated (Gastrointestinal disorders) | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 1
Cardiac failure (Cardiac disorders) | 0 | 1
Cardiac failure congestive (Cardiac disorders) | 0 | 4
Chest pain (General disorders) | 1 | 2
Coagulopathy (Blood and lymphatic system disorders) | 1 | 0
Colitis (Gastrointestinal disorders) | 1 | 0
Diverticulitis (Infections and infestations) | 1 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 7 | 5
Hypertension (Vascular disorders) | 1 | 1
Hypotension (Vascular disorders) | 1 | 0
Ileus (Gastrointestinal disorders) | 1 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 1
Pericardial effusion (Cardiac disorders) | 0 | 1
Perirectal abscess (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 1 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Pyrexia (General disorders) | 2 | 0
Sepsis (Infections and infestations) | 2 | 0
Sinusitis (Infections and infestations) | 1 | 0
Wound infection (Infections and infestations) | 1 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 0
Hypovolaemia (Metabolism and nutrition disorders) | 1 | 0
Wound dehiscence (Injury, poisoning and procedural complications) | 1 | 1
Skin reaction (Skin and subcutaneous tissue disorders) | 1 | 0
Cellulitis (Infections and infestations) | 1 | 1
Appendicitis (Infections and infestations) | 1 | 0
Breast cellulitis (Infections and infestations) | 0 | 1
Catheter related infection (Infections and infestations) | 0 | 1
Catheter site cellulitis (Infections and infestations) | 1 | 0
Gastroenteritis (Infections and infestations) | 0 | 1
Postoperative wound infection (Infections and infestations) | 0 | 1
Staphylococcal sepsis (Infections and infestations) | 1 | 0
Urinary tract infection (Infections and infestations) | 0 | 1
Pancytopenia (Blood and lymphatic system disorders) | 2 | 0
Non-cardiac chest pain (General disorders) | 1 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Abdominal pain upper (Gastrointestinal disorders) | 1 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1
Oesophagitis ulcerative (Gastrointestinal disorders) | 0 | 1
Syncope (Nervous system disorders) | 1 | 2
Cerebrovascular accident (Nervous system disorders) | 1 | 0
Encephalopathy (Nervous system disorders) | 0 | 1
Deep vein thrombosis (Vascular disorders) | 2 | 0
Bone pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 1
Hepatic enzyme increased (Investigations) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | AC --> ABI-007 (N=98) | AC --> Taxol (N=99)
Nausea (Gastrointestinal disorders) | 77 | 79
Constipation (Gastrointestinal disorders) | 47 | 40
Diarrhoea (Gastrointestinal disorders) | 35 | 35
Vomiting (Gastrointestinal disorders) | 38 | 29
Stomatitis (Gastrointestinal disorders) | 17 | 27
Abdominal pain (Gastrointestinal disorders) | 16 | 9
Abdominal pain upper (Gastrointestinal disorders) | 9 | 4
Fatigue (General disorders) | 81 | 77
Mucosal inflammation (General disorders) | 37 | 30
Pyrexia (General disorders) | 21 | 25
Oedema peripheral (General disorders) | 12 | 14
Chest pain (General disorders) | 7 | 8
Asthenia (General disorders) | 11 | 6
Headache (Nervous system disorders) | 42 | 41
Neuropathy (Nervous system disorders) | 39 | 38
Neuropathy peripheral (Nervous system disorders) | 30 | 24
Dysgeusia (Nervous system disorders) | 17 | 22
Peripheral sensory neuropathy (Nervous system disorders) | 19 | 18
Dizziness (Nervous system disorders) | 17 | 16
Paraesthesia (Nervous system disorders) | 6 | 9
Alopecia (Skin and subcutaneous tissue disorders) | 61 | 66
Rash (Skin and subcutaneous tissue disorders) | 28 | 22
Nail disorder (Skin and subcutaneous tissue disorders) | 28 | 20
Erythema (Skin and subcutaneous tissue disorders) | 8 | 12
Dry skin (Skin and subcutaneous tissue disorders) | 6 | 11
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 4 | 13
Pruritus (Skin and subcutaneous tissue disorders) | 8 | 8
Arthralgia (Musculoskeletal and connective tissue disorders) | 54 | 48
Myalgia (Musculoskeletal and connective tissue disorders) | 45 | 41
Pain in extremity (Musculoskeletal and connective tissue disorders) | 26 | 27
Bone pain (Musculoskeletal and connective tissue disorders) | 14 | 14
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 45 | 38
Cough (Respiratory, thoracic and mediastinal disorders) | 27 | 37
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 23 | 25
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 16 | 20
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 15 | 12
Upper respiratory tract infection (Infections and infestations) | 24 | 15
Urinary tract infection (Infections and infestations) | 13 | 16
Hot flush (Vascular disorders) | 33 | 30
Hypertension (Vascular disorders) | 27 | 33
Anaemia (Blood and lymphatic system disorders) | 50 | 44
Neutropenia (Blood and lymphatic system disorders) | 29 | 24
Leukopenia (Blood and lymphatic system disorders) | 13 | 14
Anorexia (Metabolism and nutrition disorders) | 26 | 20
Dehydration (Metabolism and nutrition disorders) | 8 | 10
Insomnia (Psychiatric disorders) | 27 | 26
Weight decreased (Investigations) | 14 | 14
Lacrimation increased (Eye disorders) | 9 | 10
Vision blurred (Eye disorders) | 9 | 7
Proteinuria (Renal and urinary disorders) | 12 | 11
Thrombocytopenia (Blood and lymphatic system disorders) | 8 | 5
Palpitations (Cardiac disorders) | 7 | 2
Ear pain (Ear and labyrinth disorders) | 5 | 2
Tinnitis (Ear and labyrinth disorders) | 2 | 5
Dry mouth (Gastrointestinal disorders) | 2 | 7
Dyspepsia (Gastrointestinal disorders) | 19 | 25
Dysphagia (Gastrointestinal disorders) | 4 | 6
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 12 | 10
Gingival bleeding (Gastrointestinal disorders) | 6 | 3
Glossodynia (Gastrointestinal disorders) | 5 | 1
Haemorrhoids (Gastrointestinal disorders) | 13 | 10
Oral pain (Gastrointestinal disorders) | 8 | 5
Rectal haemorrhage (Gastrointestinal disorders) | 8 | 3
Catheter site pain (General disorders) | 5 | 1
Chills (General disorders) | 8 | 4
Pain (General disorders) | 7 | 7
Tenderness (General disorders) | 5 | 1
Seasonal allergy (Immune system disorders) | 3 | 5
Fungal infection (Infections and infestations) | 6 | 0
Nasopharyngitis (Infections and infestations) | 5 | 6
Pharyngitis (Infections and infestations) | 5 | 2
Rhinitis (Infections and infestations) | 8 | 4
Sinusitis (Infections and infestations) | 11 | 11
Bloody airway discharge (Injury, poisoning and procedural complications) | 5 | 4
Contusion (Injury, poisoning and procedural complications) | 5 | 0
Radiation skin injury (Injury, poisoning and procedural complications) | 11 | 6
Decreased appetite (Metabolism and nutrition disorders) | 6 | 9
Hypokalaemia (Metabolism and nutrition disorders) | 6 | 3
Back pain (Musculoskeletal and connective tissue disorders) | 11 | 16
Chest wall pain (Musculoskeletal and connective tissue disorders) | 6 | 6
Muscle spasms (Musculoskeletal and connective tissue disorders) | 5 | 4
Neck pain (Musculoskeletal and connective tissue disorders) | 3 | 5
Pain in jaw (Musculoskeletal and connective tissue disorders) | 5 | 2
Shoulder pain (Musculoskeletal and connective tissue disorders) | 5 | 9
Amnesia (Nervous system disorders) | 1 | 5
Hypoaesthesia (Nervous system disorders) | 6 | 5
Migraine (Nervous system disorders) | 1 | 5
Sinus headache (Nervous system disorders) | 2 | 5
Anxiety (Psychiatric disorders) | 10 | 15
Depression (Psychiatric disorders) | 10 | 13
Dysuria (Renal and urinary disorders) | 4 | 8
Breast pain (Reproductive system and breast disorders) | 3 | 7
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 10 | 9
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 8 | 5
Postnasal drip (Respiratory, thoracic and mediastinal disorders) | 1 | 5
Respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 5 | 4
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 | 9
Blister (Skin and subcutaneous tissue disorders) | 3 | 5
Nail discolouration (Skin and subcutaneous tissue disorders) | 5 | 2
Night sweats (Skin and subcutaneous tissue disorders) | 6 | 2
Palmar-Plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 10 | 7
Skin exfoliation (Skin and subcutaneous tissue disorders) | 4 | 5
Flushing (Vascular disorders) | 5 | 2
Lymphoedema (Vascular disorders) | 5 | 7
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 3 | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Results from a center cannot be submitted for publication before results of multicenter study are published unless it has been more than 2 years since study completion. Then, Investigator can publish if manuscript is submitted to Celgene 60 days prior to submission. If Celgene decided publication would hinder patent applications, Investigator must delay submission for up to 1 year. Investigator must delete confidential information before submission.